CLINICAL TRIAL: NCT06032078
Title: Evaluation of the Responsiveness of Investigator Global Assessment Score for Keratosis
Brief Title: Evaluation of the Responsiveness of Investigator Global Assessment Score for Keratosis Pilaris
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Premier Specialists, Australia (Other)
Collaborators: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Dedee Murrell, Professor Dedee Murrell, Premier Specialists, Australia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-04-376-A-3
Record Dates: First submitted 2023-08-28; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Keratosis Pilaris
Keywords: responsiveness; investigator global assessment
MeSH Terms: conditions — Burnett Schwartz Berberian syndrome

STUDY DESIGN:
Intervention Model Description: 15 patients with keratosis pilaris (including subtypes) are recruited
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with keratosis pilaris (Experimental): Patients treated with 3 sessions of 1064nm Nd: YAG laser at 4-weekly intervals. Results are compared with baseline.
  Interventions: Device: Cutera laser machine

INTERVENTIONS:
Device: Cutera laser machine — 1064nm Nd: YAG laser

SUMMARY:
This prospective study aims to evaluate the responsiveness of the validated investigator global assessment (IGA) and composite area index score for keratosis pilaris by data collection through treatment and scoring sessions held at a private practice and relevant statistical analysis.

DETAILED DESCRIPTION:
This is a prospective study aiming to evaluate the responsiveness of the IGA score for KP. KPAI is a 5-point IGA score (0-4) of five main body areas: face, upper limbs, lower limbs, trunk, and buttocks, for a maximum of 20 in two main categories, activity (erythema, skin roughness and papulation) and damage (pigmentation and scarring). The final score will be a maximum of 100. KPIGA, on the other hand, is a standard 0-4 IGA score. A Physician's Global Assessment Score and a 15-point Likert Scale would also be used by investigators, data collected act as external anchor for further responsiveness statistical analysis purpose.

4 scoring sessions will take place at Premier Specialists, Kogarah, Sydney with all co-investigators conducting the study in person at this single study site. Each dermatologist and medical professional involved will receive training on using the scores through a slideshow of training photos prior to the live scoring session. Firstly, a baseline score will be determined using the proposed scoring systems on the first scoring session. After that, participants will be offered 3 sessions of Nd: YAG laser 1064nm treatments at 4-week intervals on the affected skin of all body regions (face, upper limbs, lower limbs, trunk, and buttocks). The baseline KPIGA and KPAI scores obtained on the first scoring visit acts as the control for this pilot study and the scores obtained in the 3 progressive visits will be compared to the baseline. According to relevant study, the recommended Nd: YAG laser 1064nm treatment regimen is 3 treatment sessions at 4-week intervals. They will be scored before subsequent treatment sessions to see if there is any improvement in their KP and if the score is responsive to change.

Every participant will also complete the DLQI questionnaire during each visit. This data will be used to provide insight of patient's subjective perceptions of KP and the psychological impact it may have on them.

ELIGIBILITY:
Inclusion Criteria:

1. All genders are allowed to participate
2. Age range: 18-80 years
3. Participants with Fitzpatrick skin type 1-3
4. Those with KP including subtypes of KP on the scored body regions (face, upper limbs, lower limbs, trunk, and buttocks)
5. Able to attend the scoring sessions
6. Participants having read and understood the PICF and are willing to participate
7. Of mature mind and able to provide informed consent
8. Able to maintain compliance with required study related procedures including completing the QOL questionnaire's

Exclusion Criteria:

1. Participants who are unwilling or unable to attend the scoring sessions
2. Those with other skin conditions overlapping the same area(s) as the KP
3. People younger than 18
4. People with darker skin i.e. Fitzpatrick skin type 4 or above
5. Those who had received any laser or dermabrasion therapy in the previous 6 months or topical treatment (keratolytic agents or corticosteroids) in the previous 1 month before the study treatment session
6. Those with a history of keloid or hypertrophic scars
7. Those being on photosensitive medications, allergic to intervention agents
8. Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2023-12-29 (Estimated); Study Completion 2023-12-29 (Estimated)

PRIMARY OUTCOMES:
KP-IGA | through study completion, an average of 1 year
  KP-IGA is a standard 0-4 IGA score.
KPAI | through study completion, an average of 1 year
  KPAI is a 5-point IGA score (0-4) of five main body areas: face, upper limbs, lower limbs, trunk, and buttocks, for a maximum of 20 in two main categories, activity (erythema, skin roughness and papulation) and damage (pigmentation and scarring). The final score will be a maximum of 100.
Likert Scale of Magnitude of CHange | through study completion, an average of 1 year
  15-point Likert scale from -7 (deterioration) to +7 (improvement)
Physician's Global Assessment | through study completion, an average of 1 year
  10-point scale form 0 to 10 showing the worst skin condition to the best

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Premier Dermatology, Sydney, New South Wales
  - Premier Specialists, Sydney, New South Wales

IPD SHARING:
Plan to Share IPD: No
All data obtained will be stored securely on-site premises and will not be articulated outside of Australia. Data obtained from patients through scoring sheets and QOL questionnaires will be transcribed as de-identifiable data in an Excel spreadsheet into a password-protected computer (only the investigators with the corresponding study codes given to each patient can identify the data for the purpose of study data analysis). The original scoring sheets and QOL questionnaires will be stored securely on-site and may only be accessed by investigators and co-investigators, as detailed in the patient consent form.